CLINICAL TRIAL: NCT02185378
Title: Effects of 1:1 Inspiratory to Expiratory Ratios on Oxygenation and Intrapulmonary Shunt Fraction During One Lung Ventilation in the Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 4-2014-0302
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Obese Patients, One Lung Ventilation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- I:E ratio 1:2 (Active Comparator): We plan to evaluate the improvement on respiratory function with different ventilation I:E ratios (1:2 vs. 1:1) during the one-lung ventilation in an obese patients.
  Interventions: Procedure: I:E ratio 1:2
- I:E ratio 1:1 (Active Comparator): The purpose of our study is to compare the effects of minimal prolonged 1:1 IE ratioventilation on respiratory mechanics and oxygenation with conventional 1:2 IE ratio ventilation during OLV in obese patients.
  Interventions: Procedure: I:E ratio 1:1

INTERVENTIONS:
Procedure: I:E ratio 1:2 — We plan to evaluate the improvement on respiratory function with different ventilation I:E ratios (1:2 vs. 1:1) during the one-lung ventilation in an obese patients.
  Arms: I:E ratio 1:2
Procedure: I:E ratio 1:1 — The purpose of our study is to compare the effects of minimal prolonged 1:1 IE ratioventilation on respiratory mechanics and oxygenation with conventional 1:2 IE ratio ventilation during OLV in obese patients.
  Arms: I:E ratio 1:1

SUMMARY:
One-lung ventilation, even in patients with healthy weight, causes an impairment in gas-exchange and respiratory mechanics. We hypothesized that oxygenation during the one-lung ventilation in obese patients would be improved by applying inverse-ratio ventilation, reducing atelectasis in the dependent lung and resulting in reduced shunt. Because of the restrictive ventilatory effects of obesity, these patients often show a decreased functional residual capacity and decreased expiratory reserve volume, leading to an overall decreased tidal volume. These reduction leads to arterial hypoxemia, V-Q mismatch and Rt to Lt shunting. There are few studies on the one lung ventilation in obese patients about this prolonged inspiratory time ventilatory method. We plan to investigate the effect of this ventilation method in obese patients during one lung ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. Above 40 years of age.
2. American Society of Anesthesiologists (ASA) Physical Status I, II, III.
3. Obesity (BMI >25 kg/ m2 )
4. thoracic surgical procedure

Exclusion Criteria:

1. severe functional liver or kidney disease
2. diagnosed HF ( NYHA class >3)
3. reduced pulmonary diffusion capacity < 80%

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Changes of the intrapulmonary shunt fraction and respiratory dynamic parameter | T1 (10min before one lung ventibation) T2 (30min after one lung ventilation started)T3 (60min after one lung ventilation started) T4 (10min after two lung ventilation)
  shunt fraction Qs/Qt = (CcO2- CaO2)/(CcO2- CvO2), CcO2 = Hgb x 1.34 x ScO2 + PcO2 x 0.003, lung compliance : Compliance= Vt / Pplat, physiologic dead space : Vd/Vt = 1.14 x (PaCO2 - PETCO2)/PaCO2- 0.005

CONTACTS AND LOCATIONS:
Overall Officials: Young Jun Oh, MD,PhD, Principal Investigator — Department of Anaesthesiology and Pain Medicine, Anaesthesia and Pain Research Institute, Yonsei University College of Medicine
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Anaesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea